CLINICAL TRIAL: NCT03013543
Title: Setmelanotide (RM-493) Phase 2 Treatment Trial in Patients With Rare Genetic Disorders of Obesity
Brief Title: Setmelanotide Phase 2 Treatment Trial in Participants With Rare Genetic Disorders of Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-014; 2017-000387-14 (EudraCT Number)
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Genetic Obesity; Obesity; Obesity Due to Melanocortin 4 Receptor Deficiency
Keywords: Pro-opiomelanocortin (POMC) deficiency obesity; LepR deficiency obesity; Smith-Magenis Syndrome; MC4R deficiency obesity; SRC1 deficiency obesity; SH2B1 deficiency obesity
MeSH Terms: conditions — Obesity; Smith-Magenis Syndrome | interventions — setmelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 16p11.2 Cohort (Experimental): Participants with chromosomal rearrangement of the p11.2 region of chromosome 16 (16p11.2) locus causing obesity received setmelanotide once daily (QD) via subcutaneous (SC) injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- AS Cohort (Experimental): Participants with Alström syndrome (AS) received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- BBS Cohort (Experimental): Participants with Bardet-Biedl syndrome (BBS) received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- MC4R Cohort (Experimental): Participants with melanocortin-4 receptor (MC4R) deficiency obesity received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- POMC/PCSK1/LEPR Heterozygous Cohort (Experimental): Participants with pro-opiomelanocortin (POMC)/proprotein convertase subtilisin/kexin type 1 (PCSK1)/leptin receptor (LEPR) heterozygous mutations received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- POMC/PCSK1/LEPR Composite Heterozygous Cohort (Experimental): Participants with POMC/PCSK1/LEPR composite heterozygous mutations received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- POMC/PCSK1/LEPR Compound Heterozygous Cohort (Experimental): Participants with POMC/PCSK1/LEPR compound heterozygous mutations received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- SH2B1 Cohort (Experimental): Participants with steroid receptor coactivator (SRC) homology 2B adapter protein 1 (SH2B1) haploinsufficiency received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- SMS Cohort (Experimental): Participants with Smith-Magenis Syndrome (SMS) received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide
- SRC1 Cohort (Experimental): Participants with steroid receptor coactivator 1 (SRC1) mutations received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — RM-493 QD SC injection
  Other Names: RM-493

SUMMARY:
The purpose of the study was to determine the effect of setmelanotide (RM-493) on weight, hunger assessments, and other factors in participants with rare genetic disorders of obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with the following genotypes and/or clinical assessment:

   1. POMC/PCSK1/LEPR heterozygous - not currently enrolling new participants
   2. POMC/PCSK1/LEPR compound heterozygous (two different mutations in gene) or homozygous deficiency obesity
   3. POMC/PCSK1/LEPR composite heterozygous (two or more mutations in two or more genes) deficiency obesity
   4. SMS
   5. SH2B1 deficiency obesity
   6. Chromosomal rearrangement of the 16p11.2 locus causing obesity
   7. Carboxypeptidase E (CPE) compound heterozygous or homozygous deficiency obesity
   8. Leptin deficiency obesity with loss of response to metreleptin
   9. SRC1 deficiency obesity
   10. MC4R deficiency obesity
2. Age 6 years and above
3. Obese, defined as Body Mass Index (BMI) ≥ 30 kilogram per meter square (kg/m^2) for participants ≥16 years of age or BMI≥ 95th percentile for age and gender for participants 6 up to 16 years of age.
4. Participant and/or parent or guardian is able to understand and comply with the requirements of the study and is able to understand and sign the written informed consent/assent
5. Female participants of childbearing potential must be confirmed non-pregnant, and agree to use contraception as outlined in the protocol.
6. Male participants with female partners of childbearing potential must agree to a double barrier method if they become sexually active during the study. Male participants must not donate sperm during and for 90 days following their participation in the study.

Key Exclusion Criteria:

1. Recent intensive (within 2 months) diet and/or exercise regimen with or without the use of weight loss agents that has resulted in > 2% weight loss.
2. Use of any medication that is approved to treat obesity within three months of first dose of study drug (e.g., orlistat, lorcaserin, phentermine-topiramate, naltrexone-bupropion).
3. Gastric bypass surgery within the previous six months or any prior gastric bypass surgery resulting in >10% weight loss durably maintained
4. Diagnosis of schizophrenia, bipolar disorder, personality disorder, major depressive disorder, or other psychiatric disorder(s)
5. Suicidal ideation, attempt or behavior
6. Clinically significant pulmonary, cardiac, or oncologic disease
7. hemoglobin A1c (HbA1c) > 9.0% at Screening
8. History of significant liver disease
9. Glomerular filtration rate (GFR) < 30 milliliter/minute (mL/min) at Screening.
10. History or close family history of melanoma or participant history of oculocutaneous albinism
11. Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions.
12. Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.
13. Participants previously enrolled in a clinical study involving setmelanotide or any previous exposure to setmelanotide.
14. Inability to comply with QD injection regimen.
15. Females who are breastfeeding or nursing.

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (57):
- United States (43):
  - Synexus Clinical Research US, Inc. - Simon Williamson Clinic, PC, Birmingham, Alabama
  - Synexus Clinical Research US, Inc. - Phoenix Southeast, Chandler, Arizona
  - Synexus Clinical Research US, Inc. - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Honor Health Research Institute, Scottsdale, Arizona
  - Axis Clinical Trials-Downtown, Los Angeles, California
  - Axis Clinical Trials Headquarters, Los Angeles, California
  - San Diego Wake Research, San Diego, California
  - Anschutz Health and Wellness Center University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Division of Endocrinology and Diabetes Children's National Hospital, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - AXIS South Florida Clinical Trials, Hialeah, Florida
  - Florida Hospital, Orlando, Florida
  - Synexus Clinical Research US, Inc. - St. Petersburg, Pinellas Park, Florida
  - Synexus Clinical Research US, Inc. - Chicago, Chicago, Illinois
  - Maine Medical Partners, Portland, Maine
  - NIH Hatfield Clinical Research Center, Bethesda, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Medicine, Ann Arbor, Michigan
  - Precision Medicine for Obesity Research: Gastroenterology & Hepatology Mayo Clinic, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - Impact Clinical Trials, Las Vegas, Nevada
  - AXIS New York Clinical Trials, Brooklyn, New York
  - University at Buffalo, Buffalo, New York
  - AXIS Clinical Trials, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Research Inc., Raleigh, North Carolina
  - Synexus Clinical Research US, Inc. - Akron, Akron, Ohio
  - Synexus Clinical Research US, Inc. - Cincinnati, Cincinnati, Ohio
  - Synexus Clinical Research US, Inc. - Columbus, Columbus, Ohio
  - Obesity Institute, Geisinger Clinic, Danville, Pennsylvania
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Synexus Clinical Research US, Inc. - Primary Care Associates, PC, Anderson, South Carolina
  - Wake Research TN, Chattanooga, Tennessee
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Synexus Clinical Research US, Inc. - Plano, Plano, Texas
  - Synexus Clinical Research US, Inc. - San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Research Institute, Seattle, Washington
  - Marshfield Clinic Research Institute, Marshfield, Wisconsin
- University of Alberta, Edmonton, Canada
- France (3):
  - Hopital Trousseau - Nutrition et Gastroentérologie, Paris
  - Hopital de la Pitié-Salpêtrière, Paris
  - Service de pédiatrie CHU de la Réunion - Hôpital Félix Guyon, Saint-Denis
- Germany (3):
  - Charité Berlin, Berlin
  - University of Leipzig, Leipzig
  - University of Ulm, Ulm
- University General Hospital of Patras, Rio, Patras, Greece
- Edmond and Lily Safra Children's Hospital, Ramat Gan, Israel
- Erasmus MC, Rotterdam, Netherlands
- Hospital Infantil Universitario Niño Jesús, Madrid, Spain
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ervin C, Norcross L, Mallya UG, Fehnel S, Mittleman RS, Webster M, Haqq AM, Haws RM. Interview-Based Patient- and Caregiver-Reported Experiences of Hunger and Improved Quality of Life with Setmelanotide Treatment in Bardet-Biedl Syndrome. Adv Ther. 2023 May;40(5):2394-2411. doi: 10.1007/s12325-023-02443-y. Epub 2023 Mar 24. PMID 36961653
- [Derived] Meyer JR, Krentz AD, Berg RL, Richardson JG, Pomeroy J, Hebbring SJ, Haws RM. Kidney failure in Bardet-Biedl syndrome. Clin Genet. 2022 Apr;101(4):429-441. doi: 10.1111/cge.14119. PMID 35112343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 218 participants screened, 213 participants were enrolled in the study.
Period: Overall Study
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Started | 19 | 4 | 10 | 49 | 33 | 5 | 27 | 22 | 12 | 32
Completed | 19 | 2 | 7 | 37 | 22 | 2 | 20 | 13 | 9 | 22
Not Completed | 0 | 2 | 3 | 12 | 11 | 3 | 7 | 9 | 3 | 10
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 5 | 6 | 2 | 3 | 1 | 0 | 4
Not completed — Withdrawal By Parent/Guardian | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 2 | 1 | 3 | 8 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Non-Compliance With Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who received at least 1 dose of study drug and had baseline weight data.
Groups:
- 16p11.2 Cohort: Participants with chromosomal rearrangement of the 16p11.2 locus causing obesity received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
- AS Cohort: Participants with AS received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
- BBS Cohort: Participants with BBS received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
- MC4R Cohort: Participants with MC4R deficiency obesity received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
- POMC/PCSK1/LEPR Heterozygous Cohort: Participants with PCSK1/LEPR heterozygous mutations received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
- SH2B1 Cohort: Participants with SH2B1 haploinsufficiency received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
- SMS Cohort: Participants with SMS received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
- SRC1 Cohort: Participants with SRC1 mutations received setmelanotide QD via SC injection for 16 weeks. All participants initiated treatment with setmelanotide (starting dose being age dependent) and the dose was escalated up to a maximum dose of 3.0 mg QD. Participants either continued setmelanotide treatment by enrolling in an extension study (RM-493-022; NCT03651765) immediately following the last dose in this study or if the extension study was not open at the current clinic site, participants continued treatment in the current study for up to 1 year, resulting in treatment duration of up to 16 months.
- Total: Total of all reporting groups
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort | Total
Number analyzed (Participants) | 19 | 4 | 10 | 49 | 33 | 5 | 27 | 22 | 12 | 32 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (14.58) | 16.0 (3.74) | 22.5 (14.71) | 22.4 (15.28) | 36.1 (17.23) | 40.4 (19.62) | 30.7 (20.16) | 33.6 (17.88) | 19.4 (8.10) | 31.3 (17.13) | 28.1 (17.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 6 | 27 | 22 | 4 | 18 | 15 | 10 | 25 | 143
  Male | 6 | 1 | 4 | 22 | 11 | 1 | 9 | 7 | 2 | 7 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 3 | 2 | 0 | 0 | 2 | 2 | 3 | 14
  Not Hispanic or Latino | 13 | 4 | 8 | 40 | 31 | 5 | 25 | 19 | 10 | 29 | 184
  Unknown or Not Reported | 5 | 0 | 1 | 6 | 0 | 0 | 2 | 1 | 0 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 3 | 5 | 1 | 0 | 5 | 1 | 6 | 23
  White | 15 | 2 | 9 | 38 | 28 | 4 | 23 | 13 | 10 | 24 | 166
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 0 | 8 | 0 | 0 | 3 | 2 | 1 | 2 | 20
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 113.62 (38.489) | 87.28 (16.360) | 128.04 (28.631) | 117.87 (32.339) | 143.04 (30.492) | 139.05 (30.957) | 122.08 (43.315) | 129.06 (39.480) | 92.48 (24.556) | 124.07 (33.717) | 122.98 (36.142)
Waist Circumference [Mean (Standard Deviation); unit: centimeters (cm)] | 116.84 (22.179) | 109.75 (14.523) | 126.20 (19.344) | 122.52 (19.697) | 137.95 (18.529) | 134.00 (19.038) | 128.52 (28.772) | 130.28 (23.029) | 110.14 (11.807) | 123.10 (21.101) | 125.63 (22.162)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥ 5% Reduction in Body Weight From Baseline After 3 Months of Setmelanotide Treatment
Time Frame: Baseline to Month 3
Population: Participants in the FAS were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 19 | 4 | 10 | 49 | 33 | 5 | 27 | 22 | 12 | 32
Participants | 6 | 3 | 7 | 7 | 10 | 0 | 14 | 8 | 1 | 9

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE (also referred to as an adverse experience) could be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. TEAEs were defined as AEs reported after dosing on Day 1.
Time Frame: From first dose up to Month 16
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 19 | 4 | 10 | 49 | 33 | 5 | 27 | 22 | 12 | 32
Participants | 19 | 4 | 10 | 49 | 33 | 5 | 27 | 21 | 12 | 29

3. Secondary Outcome: Change From Baseline in Body Weight After 3 Months of Setmelanotide Treatment
Time Frame: Baseline, Month 3
Population: Participants in the FAS were analyzed.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 19 | 4 | 10 | 49 | 33 | 5 | 27 | 22 | 12 | 32
kg | -2.58 (4.886) | -5.16 (3.860) | -4.61 (7.771) | -1.26 (4.851) | -4.74 (7.689) | -0.11 (2.432) | -7.24 (6.657) | -3.98 (5.164) | -0.14 (2.805) | -3.96 (4.370)

4. Secondary Outcome: Percent Change From Baseline in Body Weight After 3 Months of Setmelanotide Treatment
Time Frame: Baseline, Month 3
Population: Participants in the FAS were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 19 | 4 | 10 | 49 | 33 | 5 | 27 | 22 | 12 | 32
percent change | -2.19 (3.685) | -6.38 (5.043) | -4.19 (5.579) | -0.75 (4.291) | -3.50 (5.817) | -0.31 (1.772) | -5.57 (5.170) | -2.92 (3.834) | -0.00 (3.651) | -3.34 (3.607)

5. Secondary Outcome: Change From Baseline in Daily Hunger Questionnaire Scores After 3 Months of Setmelanotide Treatment in Participants Aged ≥ 12 Years
Description: The mean change in daily hunger questionnaire scores for participants ≥ 12 years of age with obesity in treatment with setmelanotide was evaluated. On the Daily Hunger Questionnaire, each of the 3 items (average hunger in the last 24 hours, most/worst hunger in the last 24 hours, and morning hunger) was assessed daily and scored separately using a numeric rating score for each from 0 to 10, with 0 = not hungry at all and 10 = hungriest possible.
Time Frame: Baseline, Month 3
Population: Participants aged ≥ 12 years in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 14 | 4 | 6 | 36 | 31 | 4 | 17 | 19 | 0 | 29
units on a scale
  Baseline: Hunger Score on Average Last 24 hours | 6.11 (2.102) | 5.07 (1.860) | 6.37 (1.719) | 5.74 (1.915) | 5.73 (2.178) | 8.07 (1.348) | 6.32 (2.062) | 6.66 (1.966) |  | 6.04 (2.049)
  Change at Month 3: Hunger Score on Average Last 24 hours: number analyzed (Participants) | 14 | 3 | 6 | 30 | 18 | 2 | 12 | 11 | 0 | 18
  Change at Month 3: Hunger Score on Average Last 24 hours | -2.57 (2.602) | -1.23 (2.739) | -3.21 (2.858) | -2.50 (2.278) | -2.71 (1.946) | -3.21 (2.525) | -3.12 (1.911) | -2.78 (2.639) |  | -2.47 (2.003)
  Baseline: Hunger Score at Most Hungry Last 24 hours | 7.23 (2.168) | 6.06 (2.185) | 7.50 (1.407) | 6.84 (1.866) | 6.95 (2.281) | 8.82 (0.936) | 7.45 (2.376) | 7.42 (1.870) |  | 6.91 (1.952)
  Change at Month 3: Hunger Score at Most Hungry Last 24 hours: number analyzed (Participants) | 14 | 3 | 6 | 30 | 18 | 2 | 12 | 11 | 0 | 18
  Change at Month 3: Hunger Score at Most Hungry Last 24 hours | -2.85 (2.561) | -2.27 (3.656) | -4.00 (2.717) | -2.91 (2.155) | -3.00 (2.264) | -4.07 (2.929) | -3.70 (2.501) | -2.68 (2.915) |  | -2.67 (2.241)
  Baseline: Hunger Score in Morning | 5.24 (2.508) | 4.98 (3.187) | 5.31 (2.705) | 3.99 (2.805) | 3.89 (2.589) | 7.04 (2.437) | 5.14 (2.537) | 4.96 (2.829) |  | 4.60 (2.924)
  Change at Month 3: Hunger Score in Morning: number analyzed (Participants) | 14 | 3 | 6 | 30 | 18 | 2 | 12 | 11 | 0 | 18
  Change at Month 3: Hunger Score in Morning | -2.34 (3.390) | -3.90 (4.195) | -3.14 (3.173) | -2.14 (2.914) | -2.85 (2.084) | -2.36 (1.111) | -3.15 (1.781) | -3.09 (1.961) |  | -1.88 (1.942)

6. Secondary Outcome: Change From Baseline in Daily Hunger Questionnaire Scores After 3 Months of Setmelanotide Treatment in Participants Aged < 12 Years
Description: The mean change in daily hunger questionnaire scores for participants < 12 years of age with obesity in treatment with setmelanotide was evaluated. Hunger was assessed daily using a Daily Hunger Questionnaire with a pictorial (smiley face) version of the Likert rating scale with scores ranged from 0 to 4, with 0 = not hungry at all and 4 = hungriest possible.
Time Frame: Baseline, Month 3
Population: Participants < 12 years of age in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 4 | 0 | 0 | 7 | 0 | 0 | 3 | 3 | 0 | 0
units on a scale
  Baseline: Hunger Right Now | 2.32 (0.741) |  |  | 2.02 (1.300) |  |  | 2.17 (1.443) | 1.87 (0.125) |  |
  Change at Month 3: Hunger Right Now: number analyzed (Participants) | 4 | 0 | 0 | 7 | 0 | 0 | 3 | 2 | 0 | 0
  Change at Month 3: Hunger Right Now | -1.57 (0.261) |  |  | -0.72 (1.346) |  |  | -1.55 (0.910) | -1.44 (0.387) |  |

7. Secondary Outcome: Number of Participants With Shifts From Baseline in Global Hunger Questionnaire Scores After 3 Months of Setmelanotide Treatment in Participants Aged ≥ 12 Years
Description: For participants ≥ 12 years of age, the following question was asked using the Global Hunger Questionnaire: Overall, how would you rate the hunger you experience now? Possible responses were: No hunger; Mild hunger; Moderate hunger; Severe hunger; and Not answered.
Time Frame: Baseline, Month 3
Population: Participants ≥ 12 years of age in the FAS with available data were analyzed.
Measure: Number; unit: participants
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 15 | 3 | 8 | 27 | 16 | 1 | 17 | 10 | 8 | 20
participants
  No hunger (Baseline) - No hunger (Month 3) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
  No hunger (Baseline) - Mild hunger (Month 3) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  No hunger (Baseline) - Moderate hunger (Month 3) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  No hunger (Baseline) - Severe hunger (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No hunger (Baseline) - Not answered (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mild hunger (Baseline) - No hunger (Month 3) | 0 | 0 | 0 | 2 | 3 | 0 | 2 | 3 | 1 | 4
  Mild hunger (Baseline) - Mild hunger (Month 3) | 1 | 2 | 2 | 5 | 0 | 0 | 4 | 0 | 1 | 5
  Mild hunger (Baseline) - Moderate hunger (Month 3) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
  Mild hunger (Baseline) - Severe hunger (Month 3) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Mild hunger (Baseline) - Not answered (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Moderate hunger (Baseline) - No hunger (Month 3) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
  Moderate hunger (Baseline) - Mild hunger (Month 3) | 4 | 0 | 4 | 4 | 5 | 1 | 4 | 3 | 1 | 3
  Moderate hunger (Baseline) - Moderate hunger (Month 3) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2
  Moderate hunger (Baseline) - Severe hunger (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Moderate hunger (Baseline) - Not answered (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe hunger (Baseline) - No hunger (Month 3) | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0
  Severe hunger (Baseline) - Mild hunger (Month 3) | 1 | 1 | 0 | 5 | 1 | 0 | 1 | 2 | 0 | 2
  Severe hunger (Baseline) - Moderate hunger (Month 3) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
  Severe hunger (Baseline) - Severe hunger (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  Severe hunger (Baseline) - Not answered (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not answered (Baseline) - No hunger (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not answered (Baseline) - Mild hunger (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not answered (Baseline) - Moderate hunger (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not answered (Baseline) - Severe hunger (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not answered (Baseline) - Not answered (Month 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Shifts From Baseline in Global Hunger Questionnaire Scores After 3 Months of Setmelanotide Treatment in Participants Aged < 12 Years
Description: For participants < 12 years of age, the following question was asked to parents or caregivers of participants using the Global Hunger Questionnaire: How hungry is your child acting now? Possible responses were: Not hungry at all; A little hungry; Moderately hungry; Extremely hungry; and Not answered.
Time Frame: Baseline, Month 3
Population: Participants < 12 years of age in the FAS with available data were analyzed.
Measure: Number; unit: participants
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 2 | 0 | 0 | 7 | 0 | 1 | 2 | 2 | 0 | 2
participants
  Not hungry at all (Baseline) - Not hungry at all (Month 3) | 0 |  |  | 1 |  | 0 | 0 | 0 |  | 0
  Not hungry at all (Baseline) - A little hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Not hungry at all (Baseline) - Moderately hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Not hungry at all (Baseline) - Extremely hungry (Month 3) | 0 |  |  | 1 |  | 0 | 0 | 0 |  | 0
  Not hungry at all (Baseline) - Not answered (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  A little hungry (Baseline) - Not hungry at all (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  A little hungry (Baseline) - A little hungry (Month 3) | 1 |  |  | 1 |  | 1 | 2 | 1 |  | 0
  A little hungry (Baseline) - Moderately hungry (Month 3) | 0 |  |  | 1 |  | 0 | 0 | 0 |  | 0
  A little hungry (Baseline) - Extremely hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  A little hungry (Baseline) - Not answered (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Moderately hungry (Baseline) - Not hungry at all (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Moderately hungry (Baseline) - A little hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Moderately hungry (Baseline) - Moderately hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 1 |  | 0
  Moderately hungry (Baseline) - Extremely hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Moderately hungry (Baseline) - Not answered (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Extremely hungry (Baseline) - Not hungry at all (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 1
  Extremely hungry (Baseline) - A little hungry (Month 3) | 1 |  |  | 2 |  | 0 | 0 | 0 |  | 1
  Extremely hungry (Baseline) - Moderately hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Extremely hungry (Baseline) - Extremely hungry (Month 3) | 0 |  |  | 1 |  | 0 | 0 | 0 |  | 0
  Extremely hungry (Baseline) - Not answered (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Not answered (Baseline) - Not hungry at all (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Not answered (Baseline) - A little hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Not answered (Baseline) - Moderately hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Not answered (Baseline) - Extremely hungry (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0
  Not answered (Baseline) - Not answered (Month 3) | 0 |  |  | 0 |  | 0 | 0 | 0 |  | 0

9. Secondary Outcome: Percent Change From Baseline in Waist Circumference After 3 Months of Setmelanotide Treatment
Description: Waist circumference (cm) was measured according to the National Heart, Lung, and Blood Institute (NHLBI) criteria. All measurements were single measures. Waist circumference was measured when participants were in fasting condition and at approximately the same time at each visit.
Time Frame: Baseline, Month 3
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
Number analyzed (Participants) | 18 | 3 | 9 | 36 | 15 | 2 | 21 | 13 | 6 | 21
percent change | -1.00 (6.250) | -6.60 (6.828) | -4.92 (7.191) | -0.61 (11.311) | -1.09 (8.250) | 5.11 (8.412) | -5.59 (6.554) | -4.91 (8.495) | -3.83 (8.543) | -2.88 (4.632)

ADVERSE EVENTS:
Time Frame: From first dose up to Month 16
Description: Participants in the Safety Analysis Set were analyzed.
Arm/Group | 16p11.2 Cohort | AS Cohort | BBS Cohort | MC4R Cohort | POMC/PCSK1/LEPR Heterozygous Cohort | POMC/PCSK1/LEPR Composite Heterozygous Cohort | POMC/PCSK1/LEPR Compound Heterozygous Cohort | SH2B1 Cohort | SMS Cohort | SRC1 Cohort
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/4 | 0/10 | 1/49 | 0/33 | 0/5 | 0/27 | 0/22 | 0/12 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/4 | 1/10 | 1/49 | 1/33 | 1/5 | 2/27 | 0/22 | 0/12 | 0/32
Other Adverse Events (participants affected / at risk) | 19/19 | 4/4 | 10/10 | 48/49 | 33/33 | 5/5 | 27/27 | 21/22 | 12/12 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 16p11.2 Cohort (N=19) | AS Cohort (N=4) | BBS Cohort (N=10) | MC4R Cohort (N=49) | POMC/PCSK1/LEPR Heterozygous Cohort (N=33) | POMC/PCSK1/LEPR Composite Heterozygous Cohort (N=5) | POMC/PCSK1/LEPR Compound Heterozygous Cohort (N=27) | SH2B1 Cohort (N=22) | SMS Cohort (N=12) | SRC1 Cohort (N=32)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotavirus Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Typical Aura Without Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 16p11.2 Cohort (N=19) | AS Cohort (N=4) | BBS Cohort (N=10) | MC4R Cohort (N=49) | POMC/PCSK1/LEPR Heterozygous Cohort (N=33) | POMC/PCSK1/LEPR Composite Heterozygous Cohort (N=5) | POMC/PCSK1/LEPR Compound Heterozygous Cohort (N=27) | SH2B1 Cohort (N=22) | SMS Cohort (N=12) | SRC1 Cohort (N=32)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 17 | 3 | 8 | 40 | 19 | 3 | 21 | 16 | 10 | 23
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 2 | 3 | 2
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Nail Pigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Skin Striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Acanthosis Nigricans (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Melanoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lipodystrophy Acquired (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Post Inflammatory Pigmentation Change (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin Depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Butterfly Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diffuse Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ingrown Hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keloid Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pityriasis Alba (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin Sensitisation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Solar Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Solar Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria Thermal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 1 | 3 | 12 | 14 | 4 | 13 | 13 | 2 | 11
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 7 | 4 | 2 | 6 | 6 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 7 | 3 | 0 | 1 | 4 | 4 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 2 | 5 | 3 | 1 | 1 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 3 | 3 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 2 | 0 | 2 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abnormal Faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coeliac Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival Hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pigmentation Lip (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth Discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Pruritus (General disorders) | 5 | 2 | 9 | 3 | 8 | 1 | 4 | 2 | 1 | 0
Injection Site Erythema (General disorders) | 4 | 0 | 6 | 4 | 8 | 2 | 4 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 1 | 3 | 11 | 1 | 7 | 4 | 0 | 4
Injection Site Induration (General disorders) | 2 | 0 | 5 | 3 | 3 | 0 | 0 | 0 | 1 | 0
Injection Site Pain (General disorders) | 1 | 0 | 2 | 4 | 2 | 1 | 2 | 1 | 0 | 0
Injection Site Oedema (General disorders) | 0 | 0 | 7 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Injection Site Bruising (General disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Haematoma (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Temperature Intolerance (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Feeling Cold (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Discolouration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Injection Site Hypertrophy (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Inflammation (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Swelling (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chest Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling Jittery (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired Healing (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Dryness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Scab (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Warmth (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 9 | 0 | 1 | 10 | 8 | 1 | 13 | 10 | 1 | 7
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 3 | 1 | 3 | 2 | 0 | 3
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Taste Disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Poor Quality Sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 3 | 5 | 0 | 2 | 2 | 3 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 3
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 3 | 2 | 0 | 1 | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asymptomatic Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial Vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Media Acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 2 | 14 | 3 | 1 | 10 | 5 | 1 | 8
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sweat Gland Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0 | 3 | 1 | 0 | 3 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Low Density Lipoprotein Increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Urine Analysis Abnormal (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Bilirubin Increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood Triglycerides Increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Culture Urine Positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sars-Cov-2 Test Positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bilirubin Conjugated Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Cholesterol Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Cholesterol Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Lactate Dehydrogenase Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Urine Present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-Reactive Protein Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulation Test Abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Forced Vital Capacity Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glucose Urine Present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
High Density Lipoprotein Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Protein Total Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thyroid Function Test Abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Total Cholesterol/Hdl Ratio Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urobilinogen Urine Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 2 | 0 | 2 | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 2 | 3 | 2 | 1 | 1 | 0 | 1
Libido Increased (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 2
Libido Decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Terminal Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Affect Lability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Behaviour Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood Altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Panic Attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychological Factor Affecting Medical Condition (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thinking Abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erection Increased (Reproductive system and breast disorders) | 2 | 0 | 0 | 7 | 2 | 0 | 2 | 4 | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Genital Hyperaesthesia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Spontaneous Penile Erection (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Breast Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast Mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Female Sexual Arousal Disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Genital Disorder Female (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital Dysaesthesia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Labia Enlarged (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 6 | 0 | 2 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 4 | 2 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Food Craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abnormal Loss Of Weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Starvation Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 5 | 0 | 1 | 2 | 0 | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White Blood Cell Disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Animal Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Anxiety (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bundle Branch Block Right (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Excessive Cerumen Production (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle Ear Effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine Abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Age-Related Macular Degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blepharal Pigmentation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye Haematoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid Exfoliation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Immunisation Reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Developmental Hip Dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract Operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03013543/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT03013543/SAP_001.pdf